CLINICAL TRIAL: NCT02145052
Title: Optimal Method of Fascial Closure in High Risk Patients Undergoing Laparotomy: A Prospective Randomized Study
Brief Title: Optimal Method of Fascial Closure in High Risk Patients Undergoing Laparotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marc A. de Moya, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-P-000393; MGH
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Fascial Closure
Keywords: Fascial closure; Interrupted suture; Running suture; Continuous suture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous suture (Active Comparator): 0 non-looped PDS using a tapered needle starting at the superior and the inferior portions of the wound. Fascia is then approximated with at least 1cm distance from the edge of the fascia and 1cm advancement. The two sutures are then knotted in the center with 8 square knots.
  Interventions: Other: Continuous suture
- Interrupted Suture (Active Comparator): Using a tapered needle, 0 non-looped PDS interrupted figure of eight suture 1cm from the edge and advancing 1cm between each suture.
  Interventions: Other: Interrupted suture

INTERVENTIONS:
Other: Continuous suture — A continuous suture is considered standard of care.
  Arms: Continuous suture
Other: Interrupted suture — Interrupted sutures are considered standard of care.
  Arms: Interrupted Suture

SUMMARY:
The primary objective of this study is to identify the optimal method of fascial closure of a laparotomy incision in high risk patients for intra-abdominal complications. The investigators hypothesize that interrupted closure is associated with decreased complication rates when compared with running/continuous closure. Secondary objectives are to determine the rate of dehiscence in continuous and interrupted suture technique, and to determine the rate of wound infection, hernia formation, and mortality associated with suture technique.

DETAILED DESCRIPTION:
Secure wound closure is an essential requirement for an uncomplicated and expedient recovery after an abdominal operation. The incidence of dehiscence ranges from 0-6% in different patient series and the associated mortality rate ranges from 10-35% [1]. Median laparotomy is the most common technique of abdominal incisions because it is simple, provides adequate exposure, is rapid to open and usually blood sparing [2]. The two common methods of fascial closure are continuous and interrupted with absorbable or non-absorbable suture. There is little debate that there is no significant difference between the two types of suture material. However, there is an ongoing debate concerning the optimal technique for closure. Both closure techniques are considered standard of care at this time.

The best method of wound closure would be one that provides adequate tensile strength to the incision until the wound is healed, approximates the tissue in a way that normal healing mechanisms can occur under optimal circumstances, remains secure even in the presence of local or systemic infection, the suture material is well tolerated on a short and long term basis, and, finally, should be done with expediency.

Previous randomized controlled trials of abdominal fascial closure have failed to determine the best technique and ideal suture [3]. Fagniez et al. randomized 3135 patients to receive continuous or interrupted sutures and further stratified them according to the type of wound: clean, clean-contaminated, and contaminated. This study looked at all patients, elective and emergent, and there was no statistically significant difference in wound dehiscence between continuous and interrupted suture technique [4]. A similar conclusion for wound dehiscence was shown by Gislason et al. where they compared 599 adults with major GI operation who received continuous or interrupted sutures [5]. In another prospective randomized trial, 571 patients were compared for continuous vs. interrupted sutures; again the dehiscence rate was not significant between the two groups [1]. The common denominator in all of these trials was the inclusion of all patients, elective as well as emergent, undergoing a laparotomy. None of the trials have compared the suture technique for patients requiring emergency laparotomy with wound dehiscence as a primary outcome. Results of these studies were often conflicting and have left many surgeons uncertain about the ideal technique for abdominal fascial closure, leave alone patients undergoing emergency surgery.

There have been no prospective randomized trials that look at the optimal method of fascial closure in high risk patients undergoing laparotomy. Through this research study, the investigators aim to determine identify the optimal method of fascial closure (interrupted vs. running/continuous suture) of a laparotomy incision in high risk patients for intra-abdominal complications

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >18 years of age, undergoing urgent laparotomy, admitted to the Division of Trauma, Emergency Surgery, and Surgical Critical Care.

Exclusion Criteria:

1. Pregnant patients
2. All elective patients
3. Patients with pre-morbid condition not expected to survive >48 hours
4. Patients unable to communicate in English
5. Patients with primary ventral hernia or recent (within 1 month) abdominal operation.
6. Patients with mesh in place
7. Trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2008-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Dehiscence | 1 year
  Dehiscence will be defined as more than 1cm horizontal defect in the fascia along the suture lines.

SECONDARY OUTCOMES:
Wound infection | 30 days
  Surgical site infections must fulfill the following criteria:
  1. Must occur within 30 days of surgery.
  2. Must involve only the skin and subcutaneous tissue.
  3. Must involve at least one of the following: a) Purulent discharge from a superficial infection; b) Organisms isolated from aseptically obtained wound culture
  4. Must involve at least one of the following signs of infection: a) Pain or tenderness; b) Localized swelling; c) Redness or heat
Incisional Hernia | 6 months, 1 year, 5 years
  Incisional hernia will be identified by following up patients at 6 months, 1 year, and 5 years post surgery.
Mortality | 30 days
  30-day mortality is a secondary end-point.

CONTACTS AND LOCATIONS:
Overall Officials: Marc A de Moya, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified data as needed